CLINICAL TRIAL: NCT03788668
Title: Role of Hyoid Suspension With Barbed Reposition Pharyngoplasty in Management of Lateral Pharyngeal Wall Collapse in Obstructive Sleep Apnea Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ezzat Mohamed Saleh, Otorhinolaryngology Specialist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hyoid suspension & BRP in OSA
Record Dates: First submitted 2018-12-26; First posted 2018-12-27 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Hyoid suspension; Barbed reposition pharyngoplasty
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Neither the pulmonologist or the phoniatracian or the surgeon who will befrom post operative sleep study, post operative nasopharyngoscopy and post operative sleep endoscopy will know the type of operation performed to the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyoid suspension with barbed reposition pharyngoplasty (Active Comparator)
  Interventions: Procedure: Hyoid suspension
- barbed reposition pharyngoplasty (No Intervention)

INTERVENTIONS:
Procedure: Hyoid suspension — Hyoid suspension will be done with barbed reposition pharyngoplasty
  Arms: Hyoid suspension with barbed reposition pharyngoplasty

SUMMARY:
Aim of the study

To determine the exact role of hyoid bone suspension surgery in splinting lateral pharyngeal wall in the era of the lateral pharyngoplasty

DETAILED DESCRIPTION:
Before recruitment of the patients, they will be subjected to detailed history taking and full ear nose throat examination. Body mass index and neck circumference will be measured. All the patients will undergo sleep study and the following parameters will be documented: Apnea hypopnea index (AHI), lowest O2 saturation index (LSO2), mean O2 saturation and percentage of sleep time with O2 saturation below 90% (CT90%). Day time sleepiness will be assessed using Epworth sleepiness score (ESS), we will use the Arabic translated version of ESS translated and validated after a multicentric study. All the patients will be examined by flexible fiber optic nasopharyngoscopy to determine the level of obstruction using Muller's maneuver. All the patients will be subjected to Drug Induced Sleep Endoscopy (DISE) to confirm the level of obstruction and the surgeon will comment on the lateral wall collapse at the level of oropharynx and hypopharynx. All the patients will be counseled about the other options of non-invasive treatment and importance of weight reduction. All the patients will sign an informed consent.

Surgical techniques:

The first step was bilateral tonsillectomy with identification and meticulous sparing of the palatoglossus and palatopharyngeus muscles; the most important trick was to spare as much as possible the mucosal covering of both anterior and posterior pillars. Two weakening or releasing partial incisions were done by a pinpoint bowie (Colorado) at the inferior (caudal) part of the palatopharyngeal muscle. A full thickness (mucosa and muscle) triangle was removed at the superolateral corner of the tonsil to obtain a wider and most squared oropharyngeal inlet. The center of the palate was marked at palatal spine also the pterygomandibular raphe in both sides were located by digital palpation and marked. We used a single barbed suture, bidirectional polydioxanone absorbable monofilament, size 0, with transition zone in the middle. One needle was introduced at the center point then passed laterally within the palate, turning around pterygomandibular raphe till it comes out at the most superior part of the raphe at one side; the thread is pulled until it hangs at the central transition zone which is a free zone present between the two directions of the thread. The needle again is re-introduced close to point of exit, passing around the pterygomandibular raphe, till it comes out into the tonsillectomy bed, then through the upper part of the palatopharyngeus muscle and comes out near to mucosa of posterior pillar not through it. The posterior pillar is entered at the junction between the upper third and the lower two-thirds. Then, again the needle is passed back through the tonsillectomy bed and then this suture will be suspended around the raphe again; a gentle traction is then applied on the thread only and no knots are taken. This leads to a stable re-positioning of the posterior pillar to more lateral and anterior location without any knot, then Marking the center of palate, pterygomandibular raphe and squaring of anterior pillars. The barbed suture around the upper part of the right raphe and it hangs at the central transition zone. c The needle is passed through the upper part of the palatopharyngeus muscle and comes out near to mucosa of posterior pillar not through it. The needle is passed through the upper pole and suspended around the raphe, pulling of barbed suture without taking of knots this stitch is repeated at least three times between raphe and muscle till the lower pole of the muscle is reached. The opposite side is done by the same way. Finally, each thread comes out at the raphe of the same side, for locking of the stitches and looseness prevention; a superficial stitch in the opposite direction is taken, and then the thread is cut while bushing the tissue downward for more traction.

Hyoid suspension (Thyro-hyoid-pexy) will be done. The hyoid suspension procedure will be performed under general anesthesia, with the patient in supine position with the neck extended. Skin marks over the mandibular margin, hyoid bone, thyroid notch and sternal notch. The skin incision followed a horizontal skin crease between the body of the hyoid bone and the thyroid notch. The incision will be carefully extended through the subcutaneous tissue and platysma muscle, as the muscle is less defined in the midline. Upper and lower subplatysmal flaps will be elevated to expose the strap muscles, which will be separated in the midline. The plane of the thyroid cartilage and the surface of the hyoid bone will be exposed and the thyrohyoid membrane was clearly defined. Vicryl 0 will be wrapped around the body of the hyoid bone on each side of the midline with a sharp needle and then directed to the thyroid lamina of the same side piercing it from the lateral to the medial surface, about ½ cm from the upper border of the cartilage. Two sutures will be performed on each side. The sutures will be tied steadily and gently,with the neck in neutral position. The wound will be closed in layers. A suction drainage will be placed for 48 hours.

Sample size:

In this prospective study, 31 patients will be included and will be randomized into two groups. Sample size calculation was done using sample size calculator software on ww.calculator.net website.

Randomization:

Patients will be randomized in two groups; Group (A) will undergo Barbed Reposition pharyngoplasty only and group (B) will under go Barbed Reposition pharyngoplasty and hyoid suspension. Simple randomization will be done by allowing the patients to choose between two sealed envelope.

Neither the pulmonologist or the phoniatricians or the surgeon who will perform post operative sleep study, post operative nasopharyngoscopy and post operative sleep endoscopy will know the type of operation performed to the patients.

Follow up:

Patients will be subjected to another sleep study, flexible fiber optic nasopharyngoscopy, drug induced sleep endoscopy and day time sleepiness evaluation using (ESS) 4 months after the surgery.

Statistical analysis:

The data will be tested for normality using the Kolmogorov-Smirnov test and for homogeneity variances prior to further statistical analysis. Chi-square and fisher exact tests will be used to compare between categorical variables. Unpaired t-test will be used to compare between continuous variables for normally distributed data and Mann Whitney U for non-normally distributed data. A two-tailed p < 0.05 will be considered statistically significant. All analyses were performed with the International Business Machines Statistical Package for the Social Sciences International Business Machines 20.0 software.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of both sexes between 18-60 years old.
2. Moderate to severe obstructive sleep apnea diagnosed by sleep study with apnea hypopnea index (AHI) > 15/h.
3. Body mass index (BMI) <35.
4. Refusing or intolerable to use continuous positive airway pressure.
5. Lateral pharyngeal wall collapse diagnosed by drug induced sleep endoscopy.
6. Patients who underwent previous tonsillectomy, adenoidectomy or previous nasal surgeries can be included.

Exclusion Criteria:

1. Patients who are unfit for surgeries.
2. Patients who are tolerable to continuous positive airway pressure.
3. Patients who underwent any palatal, pharyngeal, oral, mandibular, maxillofacial surgeries.
4. Patients with central sleep apnea and neurological syndromes.
5. Patients with neck, cervical vertebral pathologies and hypothyroidism.
6. Patients who had facial skeletal abnormalities.
7. Patients who had kissing tonsils or adenoids or huge tongue base.
8. Patients who have other level of obstruction (beside oropharyngeal lateral wall collapse and hypopharyngeal retro lingual obstruction) will be excluded or have this level of obstruction completely managed before recruitment in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Apnea hypopnea index (AHI) | 4 months after intervention
  Number of apneas and hypopneas recorded during sleep is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation.
  Minimal: AHI < 5 per hour Mild: AHI ≥ 5, but < 15 per hour Moderate: AHI ≥ 15, but < 30 per hour Severe: AHI ≥ 30 per hour decrease in the AHI indicate better outcome
lowest O2 saturation index (LSO2) | 4 months after intervention
  Lowest 02 saturation during sleep Increase of this parameter indicate better outcome
mean O2 saturation | 4 months after intervention
  Increase this parameter indicate better outcome
percentage of sleep time with O2 saturation below 90% (CT90%) | 4 months after intervention
  Decrease in this parameter indicate better outcome
Degree of airway obstruction with Drug Induced Sleep Endoscopy (DISE) | 4 months after intervention
  Degree of obstruction will be evaluated using grading system Grade 1 (0-25%) of airway is obstructed Grade 2 (25-50%) of airway obstructed Grade 3 (50-75%) of airway is obstructed Grade 4 (75-100%) of airway is obstructed Decrease in this parameter indicate better outcome

SECONDARY OUTCOMES:
Day time sleepiness will be assessed using Epworth sleepiness score (ESS) | 4 months after intervention
  Decrease in this parameter indicate better outcome it is a questionnaire to assess the sleepniess during day time by assessment the chance of dozing during different daily activities it contain 8 question each one will be answered using a scale from 0-3 0= no dozing
  1. slight chance of dozing
  2. moderate chance of dozing
  3. high chance of dozing Total score can range from 0-24 0-5 Lower Normal Daytime Sleepiness 6-10 Higher Normal Daytime Sleepiness 11-12 Mild Excessive Daytime Sleepiness 13-15 Moderate Excessive Daytime Sleepiness 16-24 Severe Excessive Daytime Sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Saleh, MSc, Principal Investigator — Otorhinolaryngology Specialist Assiut University Hospital
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided